CLINICAL TRIAL: NCT04408924
Title: CYCLONE 1: A Phase 2 Study of Abemaciclib in Metastatic Castration-Resistant Prostate Cancer Patients Previously Treated With a Novel Hormonal Agent and Taxane-based Chemotherapy
Brief Title: Abemaciclib (LY2835219) in Men With Heavily Treated Metastatic Castration-Resistant Prostate Cancer
Acronym: CYCLONE 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17583; I3Y-MC-JPCY (Other: Eli Lilly and Company); 2020-000290-24 (EudraCT Number)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2020-05-28; First posted 2020-05-29 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: mCRPC; CDK4; CDK6; CDK4/6; CDK4&6 inhibitor; CDK4/6 inhibitor; LY2835219; CYCLONE 1; CYCLONE1
MeSH Terms: interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 200 milligram (mg) Abemaciclib Twice Daily (Experimental): Participants received 200 mg abemaciclib administered orally twice daily on a continuous dosing schedule (28-day cycle) until symptomatic and/or radiographic progression, unacceptable toxicity, or until another discontinuation criterion is met.
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219

SUMMARY:
The study will evaluate how safe and effective abemaciclib is when given to participants whose metastatic prostate cancer progresses after they had received several previous treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have metastatic prostate cancer for which castration (medical or surgical) is no longer effective (castration-resistant).
* Participant must have disease spread to soft tissue that is measurable.
* Participant must have documented evidence of progressive disease by PSA test or imaging.
* Participant must have previously received at least one of the following treatment: abiraterone acetate, apalutamide, darolutamide or enzalutamide.
* Participant must have previously received chemotherapy with docetaxel and cabazitaxel.
* Participant must be willing and amenable to undergo a biopsy of tumor tissue (or able to provide adequate archived tumor tissue sample) and to provide blood for research.
* Participant must have good physical functioning ability and adequate organ function.

Exclusion Criteria:

* Participant must not have received more than 3 therapy regimens for metastatic castration-resistant prostate cancer (NOTE: GnRHa, first-generation antiandrogens (flutamide, nilutamide, or bicalutamide), diethylstilbestrol (DES) (or other estrogens), corticosteroids, ketoconazole, and bone loss-prevention will not count as systemic therapy regimens.
* Participants must not have previously received abemaciclib or any cyclin-dependent kinase (CDK)4 and/or CDK6 inhibitors.
* Participants must not have serious and/or uncontrolled preexisting medical condition(s) including but not limited to severe renal impairment, severe hepatic impairment, interstitial lung disease (ILD)/pneumonitis, severe dyspnea at rest or requiring oxygen therapy or other serious preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study.
* Participants must not have, or suspected to have, brain metastasis.
* Participants must not have untreated spinal cord compression, evidence of spinal metastases with risk of spinal compression or structurally unstable bone lesions suggesting impending fracture.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2023-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- United States (2):
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
- France (5):
  - Centre Leon Berard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Hopital Europeen Georges Pompidou, Paris
  - Institut Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif
- Spain (7):
  - Institut Catala d'Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Corporacion Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Abemaciclib (LY2835219) in Men With Heavily Treated Metastatic Castration-Resistant Prostate Cancer (CYCLONE 1) — https://trials.lillytrialguide.com/en-US/trial/5ARvCmtBk1XeifKLCEUPWB

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 200 Milligram (mg) Abemaciclib Twice Daily
Started | 44
Received at Least One Dose of Study Drug | 44
Completed | 31
Not Completed | 13
Not completed — Off Treatment on Post-Treatment-Discontinuation Follow-up | 3
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 5
Not completed — Sponsor Decision | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of the study drug.
Groups:
- 200 mg Abemaciclib Twice Daily: Participants received 200 mg abemaciclib administered orally twice daily on a continuous dosing schedule (28-day cycle) until symptomatic and/or radiographic progression, unacceptable toxicity, or until another discontinuation criterion is met.
Arm/Group | 200 mg Abemaciclib Twice Daily
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 14
Region of Enrollment [Number; unit: participants]
  France | 14
  Spain | 27
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Objective Response (Objective Response Rate [ORR])
Description: ORR is defined as the percentage of participants with a confirmed complete response (CR) or confirmed partial response (PR) in soft tissue per response evaluation criteria in solid tumors (RECIST) version 1.1 and do not have concurrent bone progression per Prostate Cancer Clinical Trials Working Group 3 (PCWG3), as assessed by the investigator.
  ORR = (participants with confirmed CR and no bone progression) + (participants with confirmed PR and no bone progression) x 100 / all treated participants.
Time Frame: From Date of First Dose until Objective Progression (Up To 12.8 Months)
Population: All participants who received at least one dose of the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 200 mg Abemaciclib Twice Daily
Number analyzed (Participants) | 44
percentage of participants | 6.8 [0.0 to 14.3]

2. Secondary Outcome: Radiographic Progression-Free Survival (rPFS)
Description: The rPFS time is measured from the date of first dose to the earliest date of investigator-assessed radiographic progression per RECIST 1.1 for soft tissue and PCWG3 criteria for bone, or death from any cause, whichever occurred first. Participants who have neither progressed nor died will be censored at the day of their last radiographic tumor assessment (if available) or date of first dose if no post initiation (i.e., postbaseline) radiographic assessment is available.
Time Frame: From Date of First Dose until Objective Progression or Death from Any Cause (Up To 12.8 Months)
Population: All participants who received at least one dose of the study drug. Participants censored = 11.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 200 mg Abemaciclib Twice Daily
Number analyzed (Participants) | 44
months | 2.7 [1.9 to 3.7]

3. Secondary Outcome: Overall Survival (OS)
Description: OS time is measured from the date of first dose to the date of death from any cause. If the participant was alive or lost to follow-up at the time of data analysis, OS data were censored on the last date the participant was known to be alive.
Time Frame: From Date of First Dose until Date of Death from Any Cause (Up To 28 Months)
Population: All participants who received at least one dose of the study drug. Participants censored = 13.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 200 mg Abemaciclib Twice Daily
Number analyzed (Participants) | 44
months | 8.38 [5.62 to 12.69]

4. Secondary Outcome: Duration of Response (DoR)
Description: DoR is measured only for confirmed responders (participants with a confirmed soft tissue best overall response of CR or PR per RECIST 1.1 no concurrent bone progression per PCWG3). It is measured from the date of first evidence of soft tissue CR or PR to the earliest date of investigator-assessed radiographic progression or death from any cause, whichever is earlier.
Time Frame: CR or PR to Disease Progression or Death Due to Any Cause (Up to 12 Months)
Population: All randomized participants who received at least one dose of the study drug and had CR or PR responses. The median was not achieved due to insufficient sample data.
Measure: Median (Full Range); unit: months
Arm/Group | 200 mg Abemaciclib Twice Daily
Number analyzed (Participants) | 3
months | NA [3.88 to 11.18] — Median was not achieved due to insufficient sample data.

5. Secondary Outcome: Percentage of Participants Achieving CR, PR or Stable Disease (SD) (Disease Control Rate [DCR])
Description: The DCR is defined as the percentage of participants with confirmed soft tissue best overall response of CR, PR, or stable disease (SD) per RECIST 1.1, and do not have concurrent bone disease progression per PCWG3.
Time Frame: From Date of First Dose until Measured Progressive Disease or Death Due to Any Cause (Up To 12.8 Months)
Population: All participants who received at least one dose of the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 200 mg Abemaciclib Twice Daily
Number analyzed (Participants) | 44
percentage of participants | 45.5 [30.7 to 60.2]

6. Secondary Outcome: Time to Prostate-Specific Antigen (PSA) Progression
Description: Time to PSA progression is defined as the time from the date of treatment initiation to the date of first observation of PSA progression. The PSA progression is defined as a greater than or equal to (>=) 25 percentage (%) increase and an absolute increase of >=2 nanogram/milliliter (ng/mL) above the nadir (or baseline value if baseline is the smallest on study), which is confirmed by a second value obtained 3 or more weeks later.
Time Frame: From Date of First Dose until Confirmed PSA Progression (Up To 12.8 Months)
Population: All participants who received at least one dose of the study drug. Participants censored = 31.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 200 mg Abemaciclib Twice Daily
Number analyzed (Participants) | 44
months | 6.5 [3.2 to NA] — The upper 95% confidence interval (CI) not achieved as there were insufficient number of events due to high censoring rate.

7. Secondary Outcome: Percentage of Participants Who Achieved Prostate-Specific Antigen (PSA) Response (PSA Response Rate)
Description: The PSA response rate is defined as the percentage of participants with a reduction in PSA level ≥50% from baseline, confirmed with a second assessment conducted at least 3 weeks later.
Time Frame: From Date of First Dose until Confirmed PSA Progression (Up To 12.8 Months)
Population: All participants who received at least one dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 200 mg Abemaciclib Twice Daily
Number analyzed (Participants) | 44
percentage of participants | 4.6

8. Secondary Outcome: Time to Symptomatic Progression
Description: Time to symptomatic progression is defined as the time from first dose to any of the following (whichever occurred earlier): 1) symptomatic skeletal event, defined as symptomatic fracture, surgery, or radiation to bone, or spinal cord compression; 2) pain progression or worsening of disease-related symptoms requiring initiation of a new systemic anticancer therapy; and 3) development of clinically significant symptoms due to locoregional tumor progression requiring surgical intervention or radiation therapy. For participants who were not known to have symptomatic progression at the time of data analysis, data were censored on the last date at which no symptomatic progression was indicated.
Time Frame: From Date of First Dose until Symptomatic Progression (Up to 12.8 Months)
Population: All participants who received at least one dose of the study drug. Participants censored = 28.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 200 mg Abemaciclib Twice Daily
Number analyzed (Participants) | 44
months | 4.1 [3.7 to NA] — Upper 95% confidence interval (CI) was not achieved due to high censoring rate.

9. Secondary Outcome: Pharmacokinetics (PK): Maximum Plasma Concentration at Steady State (Cmax,ss) of Abemaciclib
Description: PK: Cmax,ss of abemaciclib is reported. The cycle length was 28 days.
Time Frame: Cycle (C) 1 Day (D) 1: Post dose; C1 D15, C2D1, C2D15, C3D1: Pre dose
Population: All participants who received at least one dose of study drug had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/ mL)
Arm/Group | 200 mg Abemaciclib Twice Daily
Number analyzed (Participants) | 43
nanogram per milliliter (ng/ mL) | 223 (47)

10. Secondary Outcome: PK: Minimum/Trough Concentration at Steady State (Cmin,ss) of Abemaciclib
Description: PK: Cmin,ss of abemaciclib is reported.
Time Frame: C1 D1: Post dose; C1 D15, C2D1, C2D15, C3D1: Pre dose
Population: All participants who received at least one dose of study drug had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 200 mg Abemaciclib Twice Daily
Number analyzed (Participants) | 43
ng/mL | 176 (37)

11. Secondary Outcome: PK: Maximum Plasma Concentration at Steady State (Cmax,ss) of Abemaciclib Metabolites (Total Active Species)
Description: PK: Cmax,ss of abemaciclib metabolites (Total Active Species) is reported.
Time Frame: C1 D1: Post dose; C1 D15, C2D1, C2D15, C3D1: Pre dose
Population: All participants who received at least one dose of study drug had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micromolar per liter (µmol/L)
Arm/Group | 200 mg Abemaciclib Twice Daily
Number analyzed (Participants) | 43
micromolar per liter (µmol/L) | 1.7 (79)

12. Secondary Outcome: PK: Minimum/Trough Concentration at Steady State (Cmin,ss) of Abemaciclib Metabolites (Total Active Species)
Description: PK: Cmin,ss of abemaciclib metabolites (Total Active Species) is reported.
Time Frame: C1 D1: Post dose; C1 D15, C2D1, C2D15, C3D1: Pre dose
Population: All participants who received at least one dose of study drug had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µmol/L
Arm/Group | 200 mg Abemaciclib Twice Daily
Number analyzed (Participants) | 43
µmol/L | 1.5 (80)

13. Secondary Outcome: Percentage of Participants With Expression of Ki-67 Proliferation Marker by Immunohistochemistry (IHC)
Description: Percentage of participants with expression of Ki-67 proliferation marker at baseline by immunohistochemistry.
  Baseline expression of the Ki-67 proliferation marker was evaluated by IHC utilizing a 20% or higher score to define high Ki-67 expression. The percentage of Ki-67 positive cells was defined by the number of non-apoptotic tumor cells with unequivocal brown nuclear staining (intensities ≥1 using a 0-3 scale) over the total number of non-apoptotic tumor cells. Unit of Measure is percentage of participants with low or high baseline Ki-67 expression.
Time Frame: Baseline
Population: All participants with evaluable tumor tissue specimens
Measure: Number; unit: Percentage of participants
Arm/Group | 200 mg Abemaciclib Twice Daily
Number analyzed (Participants) | 31
Percentage of participants
  Low baseline Ki-67 expression | 25.8
  High baseline Ki-67 expression | 74.2

ADVERSE EVENTS:
Time Frame: Baseline Up to 28 Months
Description: All participants who received at least one dose of the study drug.
Arm/Group | 200 mg Abemaciclib Twice Daily
All-Cause Mortality (participants affected / at risk) | 31/44
Serious Adverse Events (participants affected / at risk) | 18/44
Other Adverse Events (participants affected / at risk) | 42/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg Abemaciclib Twice Daily (N=44)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Haemoperitoneum (Gastrointestinal disorders) | 1 (2)
General physical health deterioration (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 3 (4)
Bacteraemia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Device occlusion (Product Issues) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg Abemaciclib Twice Daily (N=44)
Anaemia (Blood and lymphatic system disorders) | 16 (17)
Neutropenia (Blood and lymphatic system disorders) | 13 (18)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 5 (7)
Constipation (Gastrointestinal disorders) | 9 (11)
Diarrhoea (Gastrointestinal disorders) | 36 (57)
Nausea (Gastrointestinal disorders) | 21 (28)
Vomiting (Gastrointestinal disorders) | 16 (19)
Asthenia (General disorders) | 24 (34)
Fatigue (General disorders) | 5 (5)
Oedema peripheral (General disorders) | 6 (6)
Pyrexia (General disorders) | 6 (6)
Urinary tract infection (Infections and infestations) | 3 (4)
Blood creatinine increased (Investigations) | 7 (9)
Neutrophil count decreased (Investigations) | 4 (4)
Platelet count decreased (Investigations) | 5 (6)
Weight decreased (Investigations) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 24 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 3 (4)
Insomnia (Psychiatric disorders) | 3 (3)
Haematuria (Renal and urinary disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/24/NCT04408924/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT04408924/SAP_001.pdf